CLINICAL TRIAL: NCT02760602
Title: A 24-Month, Phase 3, Multicenter, Placebo-Controlled Study of Efficacy and Safety of Solanezumab Versus Placebo in Prodromal Alzheimer's Disease
Brief Title: A Study of Solanezumab (LY2062430) in Participants With Prodromal Alzheimer's Disease
Acronym: ExpeditionPRO
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Insufficient scientific evidence that solanezumab would likely demonstrate a meaningful benefit to participants with prodromal AD as defined by study protocol.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16349; H8A-MC-LZBE (Other: Eli Lilly and Company); 2016-000108-27 (EudraCT Number)
Record Dates: First submitted 2016-05-02; First posted 2016-05-03 (Estimated); Results first posted 2018-07-24 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-09

CONDITIONS: Alzheimer's Disease
Keywords: anti-amyloid; monoclonal antibody
MeSH Terms: conditions — Alzheimer Disease | interventions — solanezumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Solanezumab (Experimental): Solanezumab given intravenously (IV) once every 4 weeks for up to 2 years.
  Interventions: Drug: Solanezumab
- Placebo (Experimental): Placebo given IV once every 4 weeks for up to 2 years.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Solanezumab — Administered IV
  Other Names: LY2062430
  Arms: Solanezumab
Drug: Placebo — Administered IV
  Arms: Placebo

SUMMARY:
The main purpose of this study is to investigate the safety and efficacy of the study drug solanezumab in participants with prodromal Alzheimer's disease (AD).

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis by the study investigator of a clinical syndrome of cognitive impairment consistent with prodromal AD per International Working Group (IWG) diagnostic criteria or mild cognitive impairment (MCI) due to AD per National Institute on Aging-Alzheimer's Association (NIA-AA) diagnostic criteria.
* Scores 17-28 on Montreal Cognitive Assessment (MoCA) at screening.
* Scores <27 on free recall cutoff score from the Free and Cued Selective Reminding Test (FCSRT) (Picture version) at screening.
* Scores ≤4 on Modified Hachinski Ischemia Scale (MHIS).
* Scores >0 on the Functional Activities Questionnaire (FAQ).
* Has a florbetapir positron emission tomography (PET) scan or cerebrospinal fluid (CSF) result at screening consistent with the presence of amyloid pathology.

Exclusion Criteria:

* Has had MRI or computerized tomography (CT) of brain within previous 2 years showing pathology that would be inconsistent with a diagnosis of AD.
* Has known allergy to humanized monoclonal antibodies.
* Has an ongoing clinically significant laboratory abnormality, as determined by the investigator.
* Has screening MRI with results showing >4 amyloid related imaging abnormalities H (ARIA-H) micro-hemorrhages or presence of ARIA-E.
* Has any contraindications for MRI studies, including claustrophobia, the presence of metal (ferromagnetic) implants, or a cardiac pacemaker that is not compatible with MRI.
* Has received treatment with a stable dose of an acetylcholinesterase (AChEI) inhibitor or memantine for less than 2 months before randomization. (If a participant has recently stopped AChEIs and/or memantine, he or she must have discontinued treatment at least 2 months before randomization.)

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-06; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (179):
- United States (96):
  - Xenoscience, Phoenix, Arizona
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - St Josephs Hospital and Medical Center, Phoenix, Arizona
  - Banner Sun Health Research Institute, Sun City, Arizona
  - Center for Neurosciences, Tucson, Arizona
  - Arizona Health Sciences Center, Tucson, Arizona
  - Parexel Early Phase Unit at Glendale, Glendale, California
  - Pacific Neuroscience Medical Group, Oxnard, California
  - Desert Valley Research, Rancho Mirage, California
  - Pacific Research Network Inc, San Diego, California
  - Sharp Mesa Vista Hospital, San Diego, California
  - California Pacific Medical Center, San Francisco, California
  - Apex Research Institute, Santa Ana, California
  - Care Access Research LLC, Santa Clarita, California
  - California Neuroscience Research, Sherman Oaks, California
  - Care Access Research, Valencia, California
  - MCB Clinical Research Centers, Colorado Springs, Colorado
  - Mile High Research Center, Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - New England Institute for Clinical Research, Stamford, Connecticut
  - Christiana Care Research Institute, Newark, Delaware
  - Brain Matters Research, Delray Beach, Florida
  - Neuropsychiatric Research Center of Southwest Florida, Fort Myers, Florida
  - Sunrise Clinical Research, Hollywood, Florida
  - Clinical Neuroscience Solutions Inc, Jacksonville, Florida
  - Miami Jewish Health Systems, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Suncoast Clinical Research, New Port Richey, Florida
  - Sensible Healthcare, Ocoee, Florida
  - Compass Research, Orlando, Florida
  - Pensacola Research Consultants, Inc., Pensacola, Florida
  - Quantum Laboratories, Pompano Beach, Florida
  - Roskamp Institute, Sarasota, Florida
  - Axiom Research, Tampa, Florida
  - Premiere Research Institute at Palm Beach Neurology, West Palm Beach, Florida
  - Atlanta Center of Medical Research, Atlanta, Georgia
  - United Osteoporosis Center, Gainesville, Georgia
  - Christie Clinic, LLC, Champaign, Illinois
  - Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - Central DuPage Hospital, Winfield, Illinois
  - Fort Wayne Neurological Center, Fort Wayne, Indiana
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Josephson Wallack Munshower Neurology, Indianapolis, Indiana
  - Cotton O'Neil Clinic, Topeka, Kansas
  - Heartland Research Associates, Wichita, Kansas
  - Baptist Health Medical Group, Lexington, Kentucky
  - Lake Charles Clinical Trials, Lake Charles, Louisiana
  - Maine Neurology, Scarborough, Maine
  - Sheppard Pratt Health System, Baltimore, Maryland
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - PharmaSite Research Inc, Baltimore, Maryland
  - ActivMed Practices & Research, Inc, Methuen, Massachusetts
  - Donald S Marks, Plymouth, Massachusetts
  - QUEST Research Institute, Farmington Hills, Michigan
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - ClinVest, Bolivar, Missouri
  - Clinical Research Professionals, Chesterfield, Missouri
  - Millenium Psychiatric Associates LLC, Creve Coeur, Missouri
  - St Lukes Hospital, Kansas City, Missouri
  - Las Vegas Medical Research, Las Vegas, Nevada
  - Healthy Perspectives Innovative Mental Health Services, PL, Nashua, New Hampshire
  - ActivMed Practices & Research, Inc, Portsmouth, New Hampshire
  - Memory Enhancement Center of America, Inc., Eatontown, New Jersey
  - Pyramid Clinical Research, Monroe, New Jersey
  - Princeton Medical Institute, Princeton, New Jersey
  - The Cognitive and Research Center of NJ, Springfield, New Jersey
  - Advanced Memory Research Institute of New Jersey, Toms River, New Jersey
  - Bio Behavioral Health, Toms River, New Jersey
  - Albany Medical College, Albany, New York
  - Richmond Behavorial Associates, Staten Island, New York
  - Alzheimer's Memory Center, Charlotte, North Carolina
  - Piedmont Medical Research, Winston-Salem, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Neurology Diagnostics, Inc., Dayton, Ohio
  - Insight Clinical Trials, Shaker Heights, Ohio
  - Summit Research Network Inc, Portland, Oregon
  - Center for Cognitive Health, Portland, Oregon
  - Abington Neurological Associates, Abington, Pennsylvania
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Lehigh Center for Clinical Research, Allentown, Pennsylvania
  - Clinical Trial Center, LLC, Psychiatry, Jenkintown, Pennsylvania
  - Northeastern Pennsylvania Memory & Alzheimer's Center, Plains, Pennsylvania
  - Rhode Island Mood & Memory Research Institute, East Providence, Rhode Island
  - Butler Hospital, Providence, Rhode Island
  - Metrolina Neurological Research Institute, Old Point Station, South Carolina
  - Baylor AT&T Memory Center, Dallas, Texas
  - FutureSearch Trials, Dallas, Texas
  - Houston Methodist, Houston, Texas
  - University of Texas Health Services Center - Houston, Houston, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Univ of Texas Health Science Center at San Antonio, San Antonio, Texas
  - The Memory Clinic, Bennington, Vermont
  - Sentara Medical Group, Norfolk, Virginia
  - National Clinical Research - Richmond, Richmond, Virginia
  - Evergreen Professional Plaza, Kirkland, Washington
  - Dean Foundation for Health Research and Education, Middleton, Wisconsin
- Canada (9):
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Gatineau
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Greenfield Park
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Halifax
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Kentville
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., London
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Ottawa
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Peterborough
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Sherbrooke
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Toronto
- Finland (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kuopio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oulu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampere
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Turku
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vaasa
- France (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Amiens
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bordeaux
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bron
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marseille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montpellier
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rennes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Strasbourg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toulouse
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chemnitz, Germany
- Italy (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Genova
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monza
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pavia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Perugia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pisa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Roma
- Japan (13):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bunkyō City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hachiōji
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kamakura
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kodaira-shi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kōriyama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kyoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mitaka-shi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shinjuku-Ku
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shizuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Takamatsu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tsu
- Poland (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bialystok
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bydgoszcz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lublin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poznan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sopot
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
- Puerto Rico (6):
  - Santa Cruz Behavioral PSC, Bayamón
  - Cortex, PSC, Las Piedras
  - University Of Puerto Rico, Rio Piedras
  - Instituto de Neurologia Dra. Ivonne Fraga, San Juan
  - Latin Clinical Trial Center, San Juan
  - SomniCare Sleep Institute, San Juan
- Spain (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Castellon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Donostia / San Sebastian
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Getafe
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Getxo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Plasencia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salt
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valencia
- Sweden (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Malmo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mölndal
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stockholm
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Umeå
- Taiwan (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Changhua
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gwei Shan Township
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kaohsiung City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taichung
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tainan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zhonghe
- United Kingdom (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bath
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chelsea
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guildford
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Manchester
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Scotland

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: Click here for more information about this study: A Study of Solanezumab (LY2062430) in Participants With Prodromal Alzheimer's Disease — http://www.lillytrialguide.com/en-US/studies/mild-cognitive%20impairment/LZBE#?postal=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized by site and by use of florbetapir positron emission tomography (PET) scanning or cerebrospinal fluid (CSF) for study eligibility.
Period: Overall Study
Arm/Group | Solanezumab | Placebo
Started | 13 | 13
Completed | 0 | 0
Not Completed | 13 | 13
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Terminated by sponsor | 12 | 13

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least one dose of study drug.
Groups:
- Solanezumab: Solanezumab given IV once every 4 weeks for up to 2 years.
- Total: Total of all reporting groups
Arm/Group | Solanezumab | Placebo | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.46 (6.01) | 75.62 (4.93) | 74.54 (5.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 9 | 7 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 13 | 25
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 1 | 1
  White | 9 | 12 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 11 | 21
  Japan | 2 | 0 | 2
  Canada | 1 | 0 | 1
  Poland | 0 | 2 | 2
ADAS-Cog14 at Baseline [Mean (Standard Deviation); unit: units on a scale] — ADAS-Cog14 is ADAS-Cog11 augmented with orientation, verbal memory, language, praxis, delayed free recall, digit cancellation, and maze-completion measures. The ADAS-Cog14 scale ranges from 0 to 90. Higher scores indicate greater disease severity.
  units on a scale | 24.08 (8.00) | 27.77 (3.63) | 25.92 (6.37)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Alzheimer´s Disease Assessment Scale- Cognitive Subscale (ADAS-Cog14) Score
Description: ADAS-Cog14 is ADAS-Cog11 augmented with orientation, verbal memory, language, praxis, delayed free recall, digit cancellation, and maze-completion measures. The ADAS-Cog14 scale ranges from 0 to 90. Higher scores indicate greater disease severity.
Time Frame: Baseline, 24 Months
Population: Zero participants were analyzed as no data collected.
Arm/Group | Solanezumab | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change From Baseline on Alzheimer´s Disease Cooperative Study-Activities of Daily Living Scale for Mild Cognitive Impairment (ADCS-MCI-ADL)
Description: The ADCS-MCI-ADL is a functional evaluation scale for MCI patients, based on information provided by an informant that describes the performance of participants in several ADLs. Total score ranges from 0 to 69; lower score indicates greater disease severity.
Time Frame: Baseline, 24 Months
Population: Zero participants were analyzed as no data collected.
Arm/Group | Solanezumab | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change From Baseline on the Mini Mental Status Examination (MMSE)
Description: MMSE is a brief screening instrument used to assess cognitive function (orientation, memory, attention, ability to name objects, follow verbal/written commands, write a sentence, and copy figures) in elderly participants.Total score ranges from 0 to 30; lower score indicates greater disease severity.
Time Frame: Baseline, 24 Months
Population: Zero participants were analyzed as no data collected.
Arm/Group | Solanezumab | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change From Baseline on the Montreal Cognitive Assessment (MoCA)
Description: The MoCA will be used as the global cognitive screening instrument. It will also be administered in the clinical trial at baseline and the final visits of each phase as a secondary outcome measure of global cognition. Scores on the MoCA range from 0-30 with 26-30 indicating normal global cognition.
Time Frame: Baseline, 24 Months
Population: Zero participants were analyzed as no data collected.
Arm/Group | Solanezumab | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change From Baseline on the Functional Activities Questionnaire (FAQ)
Description: FAQ is a 10-item, caregiver-based questionnaire and was administered to the study partner who was asked to rate the participant's ability to perform a variety of activities ranging from Writing checks, Assembling tax records, shopping, playing games, food preparation, traveling, keeping appointments, Traveling out of neighborhood, keeping track of current events and understanding media. FAQ total score was calculated by adding the scores from each of the 10 items. Each activity is rated on a scale from 0 to 3 (Never did and would have difficulty now = 1; Never did [the activity] but could do now = 0; Normal = 0; Has difficulty but does by self = 1; Requires assistance = 2; Dependent = 3). The maximum FAQ total score is 30, with higher scores indicating greater impairment.
Time Frame: Baseline, 24 Months
Population: Zero participants were analyzed as no data collected.
Arm/Group | Solanezumab | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change From Baseline on the Neuropsychiatric Inventory (NPI)
Description: The NPI is a tool for assessing psychopathology in participants with dementia and other neurologic disorders. Information is obtained from a caregiver familiar with the participant's behavior. The score ranges from 12 to 144, with higher scores indicating greater disease severity.
Time Frame: Baseline, 24 Months
Population: Zero participants were analyzed as no data collected.
Arm/Group | Solanezumab | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change From Baseline on the Clinical Dementia Rating Scale Sum of Boxes (CDR-SB)
Description: CDR-SB is a semi-structured interview of participants and their caregivers. Participant's cognitive status is rated across 6 domains of functioning, including memory, orientation, judgment/problem solving, community affairs, home/hobbies, and personal care. Severity score assigned for each of 6 domains; total score (SB) ranges from 0 to 18. Higher scores indicate greater disease severity.
Time Frame: Baseline, 24 Months
Population: Zero participants were analyzed as no data collected.
Arm/Group | Solanezumab | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change From Baseline on the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS)
Description: RBANS is a brief neurocognitive battery with four alternate forms, measuring immediate and delayed memory, attention, language, and visuospatial/constructional skills.
Time Frame: Baseline, 24 Months
Population: Zero participants were analyzed as no data collected.
Arm/Group | Solanezumab | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change From Baseline on the Free and Cued Selective Reminding Test (FCSRT)
Description: The FCSRT is a neuropsychological test of memory under conditions that control attention and cognitive processing in order to obtain an assessment of memory unconfounded by normal age-related changes in cognition.
Time Frame: Baseline, 24 Months
Population: Zero participants were analyzed as no data collected.
Arm/Group | Solanezumab | Placebo
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change From Baseline on the Resource Utilization in Dementia-Lite (RUD-Lite)
Description: RUD-Lite assesses the healthcare resource utilization of participants and their caregivers to determine the level of formal and informal care attributable to Alzheimer's Disease (AD). Information on both caregivers (caregiving time, work status) and participants (accommodation and healthcare resource utilization) is collected from the baseline and follow-up interviews.
Time Frame: Baseline, 24 Months
Population: Zero participants were analyzed as no data collected.
Arm/Group | Solanezumab | Placebo
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Change From Baseline on the EuroQol 5-Dimensional Health-Related Quality of Life Scale (EQ-5D)
Description: EQ-5D (proxy version) measures mobility, self-care, usual activities, pain/discomfort, anxiety/depression; each has 3 severity levels (no, some, severe problems) coded to a 1-digit number (1-3). Digits are combined into 5-digit number describing health state. Visual analogue scale (VAS) assesses caregiver's impression of participant's overall health state; scores range: 0 to 100. Lower scores indicate greater disease severity.
Time Frame: Baseline, 24 Months
Population: Zero participants were analyzed as no data collected.
Arm/Group | Solanezumab | Placebo
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Change From Baseline on the Quality of Life in Alzheimer's Disease Scale (QoL-AD)
Description: QoL for AD assess participant rates mood, relationships, memory, finances, physical condition, and overall QoL assessment. Each of 13 items rated on a 4-point scale. Sum of items=total score (range: 13-52). Higher scores=greater QoL.
Time Frame: Baseline, 24 Months
Population: Zero participants were analyzed as no data collected.
Arm/Group | Solanezumab | Placebo
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Change From Baseline in Concentration of Plasma Amyloid-β Peptide (Aβ) and Plasma Solanezumab
Description: Concentration of amino acid peptide known as Aβ 1-42 in plasma.
Time Frame: Baseline, 24 Months
Population: Zero participants were analyzed as no data collected.
Arm/Group | Solanezumab | Placebo
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Change From Baseline in Volumetric Magnetic Resonance Imaging (vMRI)
Description: MRI will be used to assess the effect of treatment on rate of whole brain volume.
Time Frame: Baseline, 24 Months
Population: Zero participants were analyzed as no data collected.
Arm/Group | Solanezumab | Placebo
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Change From Baseline in Florbetapir Positron Emission Tomography (PET) Standardized Uptake Value Ratio (SUVr)
Description: Florbetapir F18 PET used to assess the treatment effect in brain amyloid plaque deposition from baseline through 18 months as measured by florbetapir F18 PET Standardized Uptake Uptake Value ratio.
Time Frame: Baseline, 24 Months
Population: Zero participants were analyzed as no data collected.
Arm/Group | Solanezumab | Placebo
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Change From Baseline in Concentration of Cerebrospinal Fluid (CSF) Aβ and CSF Tau Proteins
Description: Changes in CSF parameters, including total and free Aβ1-40 and Aβ1-42 species and total tau and P-tau181 peptides, will be assessed.
Time Frame: Baseline, 24 Months
Population: Zero participants were analyzed as no data collected.
Arm/Group | Solanezumab | Placebo
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Change From Baseline in Neocortical Tau Deposits Using 18F-AV-1451 PET
Description: Biomarker change will be analyzed to provide biomarker-based evidence that solanezumab affects the underlying disease pathology.
Time Frame: Baseline, 24 Months
Population: Zero participants were analyzed as no data collected.
Arm/Group | Solanezumab | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline to Study Termination (Up To 11 Months)
Arm/Group | Solanezumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 2/13 | 1/13
Other Adverse Events (participants affected / at risk) | 7/13 | 1/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Solanezumab (N=13) | Placebo (N=13)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Solanezumab (N=13) | Placebo (N=13)
Coronary artery disease (Cardiac disorders) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Extravasation (General disorders) | 1 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (4) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Endodontic procedure (Surgical and medical procedures) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated due to insufficient scientific evidence that solanezumab would likely demonstrate a meaningful benefit to pts with prodromal AD as defined by the study protocol. Zero pts were analyzed as no data collected for outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2016-03-28): https://cdn.clinicaltrials.gov/large-docs/02/NCT02760602/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-08): https://cdn.clinicaltrials.gov/large-docs/02/NCT02760602/SAP_001.pdf